CLINICAL TRIAL: NCT02322086
Title: A Phase 2 Study of Cellular and Immunologic Changes in the Skin of Subjects Receiving PH-10 Aqueous Hydrogel to Plaque Psoriasis
Brief Title: A Phase 2 Study of Cellular and Immunologic Changes in the Skin of Subjects Receiving PH-10
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Provectus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-10-PS-24
Record Dates: First submitted 2014-12-16; First posted 2014-12-22 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Rose Bengal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PH-10 (Experimental): Active treatment
  Interventions: Drug: Topical Rose Bengal, 0.005%

INTERVENTIONS:
Drug: Topical Rose Bengal, 0.005% — Subjects will apply PH-10 vehicle daily for 28 consecutive days followed by active PH-10 daily for 28 consecutive days to their plaque psoriasis areas on the trunk or extremities (excluding palms, soles, scalp, facial and intertriginous sites).
  Other Names: PH-10

SUMMARY:
This is a multicenter study of subjects with mild to moderate psoriasis. Subjects will apply PH-10 vehicle daily for 28 consecutive days followed by active PH-10 daily for 28 consecutive days to their plaque psoriasis areas on the trunk or extremities (excluding palms, soles, scalp, facial and intertriginous sites). Biopsies of one target plaque will be collected at baseline (at least 7 days prior to first study treatment on Day 1) and at Days 29 and 64, with a 7-day interval between biopsy at Day 29 and commencement of application of application of active PH-10 on Day 36. Study data from each subject will serve as an internal control (i.e., assessment at baseline and at the end of application of PH-10 vehicle) for assessment of clinical and cellular response to active investigational agent.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, age 18 or older.
* Presence of mild to moderate plaque psoriasis on the trunk or extremities (excluding palms, soles, scalp, and facial or intertriginous areas).
* At least one target plaque having a minimum diameter of 5 cm (2 inches) with uniform mild to moderate plaque psoriasis.
* Fitzpatrick skin type I-VI.
* Written informed consent by the subject or legal guardian.

Exclusion Criteria:

* Female subjects of childbearing potential who are pregnant, attempting to conceive, not using effective contraception, or who are nursing an infant.
* Subjects who have received PH-10.
* Subjects who have received PUVA or systemic antipsoriatic therapy (immunosuppressants, cytostatics, corticosteroids) within 28 days of study initiation (14 days for methotrexate).
* Subjects who have received UVB light therapy within 14 days of study initiation.
* Subjects who have received topical antipsoriatic therapy (including corticosteroids, tar, anthralin or Vitamin D analogs) to the study plaque areas within 14 days of study initiation.
* Subjects who have received any approved or investigational biologic drug therapy for psoriasis within 90 days or 5 half-lives of study initiation.
* Subjects who have participated in a clinical research study within 28 days of study initiation.
* Subjects with a history of porphyria, systemic lupus erythematosus or xeroderma pigmentosum.
* Subjects with clinical conditions that, in the opinion of the Investigator, may pose a health risk to the subject because of involvement in the study or detrimentally affect regular follow-up of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in the immunologic, structural and hyperproliferative state of the skin in the target plaque and evidence of cellular atypia following PH-10 application | 28 days

SECONDARY OUTCOMES:
Psoriasis Severity Index (PSI) changes from pre-treatment | 28 days
Plaque Response changes from Day 1 pre-treatment | 28 days
Pruritus Self-Assessment score changes from Day 1 pre-treatment | 28 days
Correlation of PSI changes with observed histopathologic and immunohistopathologic changes in the skin of the target plaque | 28 days
Incidence of adverse experiences | 28 days
Incidence of adverse changes in clinical laboratory tests | 28 days
Incidence of adverse changes in weight or vital signs | 28 days
Correlation of adverse experiences with observed histopathologic and immunohistopathologic changes in the skin | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wachter, Ph.D., Study Director — Provectus Biopharmaceuticals, Inc.
Locations (3):
- United States (3):
  - International Dermatology Research, Miami, Florida
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina
  - DermResearch Inc., Austin, Texas